CLINICAL TRIAL: NCT06705062
Title: A Multi-center Randomized Clinical Study Comparing Reduced-dose (35mg/kg) Versus Standard Dose (50mg/kg) Post-transplantation Cyclophosphamide in Combination with Post-engraftment Anti-thymoglobin (ATG) and Tacrolimus and Post-engraftment Anti-thymoglobin As Graft Versus Host Disease (GVHD) Prophylaxis in Patients Undergo Alternative Donor Peripheral Hematopoietic Stem Cell Transplantation
Brief Title: Study Comparing Reduced Versus Standard Dose Post-transplantation Cyclophosphamide in Combination with Post-engraftment Anti-thymoglobin As Graft Versus Host Disease Prophylaxis in Alternative Donor Peripheral Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PTCY-REDSTAR-2024
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Allogeneic Hematopoietic Cell Transplant; Graft Versus Host Disease
Keywords: post-transplantation cyclophosphamide; prophylaxis; reduced dose; graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced dose of post-transplantation cyclophosphamide (Experimental): study group
  Interventions: Drug: reduced-dose PTCy
- Standard-dose PTCy (Active Comparator): Patients receiving standard dose of post-transplantation cyclophosphamide
  Interventions: Drug: Standard dose PTCY

INTERVENTIONS:
Drug: reduced-dose PTCy — Patients receiving reduced dose of PTCy at 35mg.kg on day +3 and +4 together with tacrolimus starting from day+5 and single dose of anti-thymoglobin (ATG) 2.5mg/kg at 72 hours after documentation of neutrophil engraftment.
  Arms: Reduced dose of post-transplantation cyclophosphamide
Drug: Standard dose PTCY — Patients receiving standard dose PTCy at 50mg/kg on day +3 and +4 with tacrolimus starting from day +5 and single dose of anti-thymoglobin at 2.5mg/kg 72 hours after documentation of neutrophil engraftment.
  Arms: Standard-dose PTCy

SUMMARY:
This is a multi-center randomized study to compare the reduced-dose of post-transplantation cyclophosphamide (PTCY) at 35mg.kg to standard dose at 50mg/kg combined with tacrolimus and post-engraftment low dose anti-thymoglobin (ATG) as graft versus host disease (GVHD) prophylaxis in patients undergoing allogeneic stem cell transplantation from alternative donor.

DETAILED DESCRIPTION:
This is a multi-center randomized study in patients undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT) from alternative donors (9-10/10 matched unrelated donor or haplo-identical donors). The aim is to evaluate to the efficacy and feasibly of reduced-dose of PTCY at 35mg/kg as GVHD prophylaxis. Patients will be assigned to study group receiving PTCy at 35mg/kg on day +3 and +4 together with tacrolimus starting from day +5 and single dose anti-thymoglobin at 2.5mg/kg as GVHD prophylaxis or to the control group with standard dose of PTCY at 50mg/kg on day +3 and +4 with same dose of tacrolimus and ATG as the study group.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergo allo-HSCT with matched unrelated donor or haplo-identical donor;
2. normal organ function (creatinine clearance ≥ 50ml/min/1.73m2 or creatinine ≤2mg/d(or 177μmol/L); no hepatic abnormal (ALT or AST≤2.5xN; TBil≤1.5XN); Normal pulmonary function (FEV1、 FVC、DLCO≥80%); normal cardiac function (EFS ≥50%);
3. ECOG: 0-2;
4. Life expectation ≥3 months;
5. Informed consent provided.

Exclusion Criteria:

1. Pregnancies
2. active hepatitis (HBV-DNA≥1×103 copies/ml);
3. active infection require anti-biotics;
4. HIV infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
100-day II-IV acute GVHD | 100 day
  Patients diagnosed with grade II-IV acute GVHD within 100 day after allo-HSCT

SECONDARY OUTCOMES:
100-day acute GVHD | 100 day
  Patients diagnosed with aGVHD of all grades within 100 days after allo-HSCT
100-day non-relapse mortality | 100 day
  Patients died of any causes without documentation of disease relapse or progression at day 100 after allo-HSCT
1-year chronic GVHD | 1 year
  Patients diagnosed with chronic GVHD of all grades at 1 year after allo-HSCT
1-year moderate to severe chronic GVHD | 1 year
  Patients diagnosed with moderate to severe chronic GVHD at 1 year after allo-HSCT
1-year NRM | 1 year
  Patients died of any causes without documentation of relapse or disease progression 1 year after allo-HSCT
1-year cumulated incidence of relapse | 1 year
  Patients died of relapse or disease progression 1 year after allo-HSCT
1-year overall survival | 1 year
  Patients remained alive at 1 year after allo-HSCT
1-year graft host disease free and relapse free survival | 1 year
  Patients remained alive without relapse, grade III-IV aGVHD or moderate to severe chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin hsopital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided